CLINICAL TRIAL: NCT00510315
Title: Abdominal Obesity and Cardiovascular Risk Factors in Women Who Survived Cancer or a Related IllnessFollowing Total Body Irradiation and Stem Cell Transplant
Brief Title: Abdominal Obesity and Cardiovascular Risk Factors in Women Who Survived Cancer or a Related Illness Following Total Body Irradiation and Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Queen's University, Kingston, Ontario (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 07-092
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Leukemia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Myelodysplastic Syndrome
Keywords: leukemia; survivors; women; leukemia survivors; cancer or a related illness; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; myelodysplastic syndrome; aplastic anemia; treated with total body irradiation; followed by an allogeneic or autologous stem cell transplant
MeSH Terms: conditions — Leukemia; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Neoplasms; Anemia, Aplastic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood

GROUPS / COHORTS (2):
- Women treated with SCT/TBI
  Interventions: Other: Questionnaires, Laboratory tests, Abdominal MRI
- 1:1 Matched group of women: Current age + or - 2 years
  Race and ethnicity
  Cancer diagnosis
  Interval from completion of cancer therapy to study + or - 2 years
  Interventions: Other: Questionnaires, Laboratory tests, Abdominal MRI

INTERVENTIONS:
Other: Questionnaires, Laboratory tests, Abdominal MRI — Height, weight, waist and hip circumference; systolic and diastolic blood pressure; questionnaires; fasting blood tests: insulin, glucose, lipids (low density lipoprotein (LDL), high density lipoprotein (HDL), triglycerides, LDL pattern, HDL and LDL subspecies), cardiac inflammatory markers (hsCRP, IL-1B, IL-6, IL-10, TNFa), leptin, adiponectin, IGF-1, and IGFBP3; abdominal MRI for visceral and subcutaneous fat measurement

SUMMARY:
The purpose of this study is to better understand why some women who survived cancer or a related illness later develop diabetes, problems with their cholesterol, or other problems that may lead to heart disease. Because these problems may be related to treatment with total body irradiation and a stem cell transplant, the investigators will compare the rates of obesity, cholesterol problems, and diabetes between women who were treated with total body irradiation and a stem cell transplant and women who were not.

The amount and location of fat stores in the abdomen is more important than overall weight or total body fat in the development of diabetes and cholesterol problems. In general, fat can be stored in several areas in the abdomen: around the organs (visceral fat), under the skin (subcutaneous fat), and in the liver (liver fat). People with higher amounts of fat around the organs (visceral fat), even those with a normal weight, are more likely to become diabetic or have high cholesterol. The amount of fat in each of these areas can be measured with an abdominal magnetic resonance imaging (MRI).

In this study, the investigators will use blood tests, height, weight, waist circumference, blood pressure measurements, and an abdominal MRI to evaluate for several risk factors of heart disease, including cholesterol problems, diabetes and pre-diabetes, elevated blood pressure, and increased abdominal fat.

DETAILED DESCRIPTION:
We will enroll 60 female participants in this study. From the population of interest, female cancer survivors (or women treated for a related illness) who were treated with TBI prior to a SCT, we will enroll 30 participants, 10 from each of the following cancer groups: acute lymphoblastic leukemia, acute myeloid leukemia, and chronic myeloid leukemia. We are interested in determining the outcomes in adult survivors who have completed their growth by the time of study and yet are younger than the age when most women generally begin to develop insulin resistance or dyslipidemia in the general population. For this reason, we will enroll women who are 18 - 49 years of age at the time of study.

ELIGIBILITY:
Inclusion Criteria:

Target population

* Females 18 - 49 years of age at time of study
* Previous diagnosis of ALL, AML, CML, CLL, Hodgkin's lymphoma, Non-hodgkin's lymphoma, aplastic anemia, and myelodysplastic syndrome
* Previously treated with TBI (1200 - 1500 cGy) prior to SCT
* Free of cancer
* Two years or more from completion of cancer therapy
* Able and willing to give informed consent

Comparison group

* Females 18 - 49 years of age at time of study
* Previous diagnosis of ALL, AML, CML CLL, Hodgkin's lymphoma, Non-hodgkin's lymphoma, aplastic anemia, and myelodysplastic syndrome
* Free of cancer
* Two years or more from completion of cancer therapy
* Able and willing to give informed consent

Exclusion Criteria:

Target population

* Pregnant at time of study
* Previous cranial radiotherapy (other than TBI)
* Second primary malignancy (other than non-melanoma skin cancer)
* Any patient who has received glucocorticoids or tacrolimus within 60 days prior to the study
* Currently on a medication for diabetes mellitus or dyslipidemia
* Patients with a creatinine > 1.5 mg/dL or biopsy-proven chronic active hepatitis
* Contraindication to an MRI

Comparison group

* pregnant at time of study
* Previous cranial radiotherapy
* Second primary malignancy (other than non-melanoma skin cancer)
* Any patient who has received glucocorticoids or tacrolimus within 60 days prior to the study
* Currently on a medication for diabetes mellitus or dyslipidemia
* Patients with a creatinine > 1.5 or biopsy-proven chronic active hepatitis
* Contraindication to an MRI

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential research subjects will be identified by a member of the research team from the SCT database and the medicine and pediatrics leukemia databases.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Explore whether visceral adipose tissue is significantly higher in women who were treated with total body irradiation (TBI) plus stem cell transplant in comparison with women who were not | within 12 months

SECONDARY OUTCOMES:
Determine the differences in processes of changes, decisional balance for physical activity, body image, mood, and quality of life between the groups | within 12 months
Determine the correlation between the amount of visceral adipose tissue and fasting levels of triglycerides, LDL, HDL, insulin, glucose, and HOMA-IR in both groups. | within 12 months
To begin to characterize the psychosocial risk factors of the TBI plus stem cell transplant group, in relation to the comparison group, in order to inform a future targeted intervention to reduce risk. | within 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Oeffinger, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Background] Oeffinger KC, Adams-Huet B, Victor RG, Church TS, Snell PG, Dunn AL, Eshelman-Kent DA, Ross R, Janiszewski PM, Turoff AJ, Brooks S, Vega GL. Insulin resistance and risk factors for cardiovascular disease in young adult survivors of childhood acute lymphoblastic leukemia. J Clin Oncol. 2009 Aug 1;27(22):3698-704. doi: 10.1200/JCO.2008.19.7251. Epub 2009 Jun 29. PMID 19564534
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org